CLINICAL TRIAL: NCT06852339
Title: Bringing Evidence to the Point-of-Care in Chronic Obstructive Pulmonary Disease: the EAPOC-COPD System
Brief Title: Evaluating the EAPOC-COPD System
Acronym: EAPOC-COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Andrew Kouri, Scientist and Staff physician, Women's College Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSI Grant Number: 24-08
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: COPD; clinical decision support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinding will not be possible for participating providers or patients, given the nature of the EAPOC-COPD intervention as a point-of-care clinical decision support system integrated into routine care workflows. However, outcome assessors conducting the chart reviews will be blinded to the intervention status of the site and the period during which data were collected to minimize the risk of bias in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EAPOC-COPD system (Experimental): The EAPOC-COPD system consists of: 1) a smart phone / tablet app or PC-based questionnaire which collects information directly from patients upon prompting, up to 1 week before their clinical appointment; and 2) a point-of-care CDSS that wirelessly receives and processes questionnaire data in order to produce a symptom severity/exacerbation risk assessment, medication change recommendation, and COPD action plan, all of which is made available to providers through a prompt, upon opening the patient chart in the existing EMR. Once approved, the personalized COPD action plan is automatically populated within the patient app/portal, enabling anywhere/anytime access for patients. Patients are also provided with educational resources within their app/portal, designed to improve health literacy, inhaler technique, and adherence to their action plan.
  Interventions: Behavioral: EAPOC-COPD
- Control arm (Active Comparator): Prior to activation of the EAPOC-COPD system, providers will provide usual care to their patients with COPD
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: EAPOC-COPD — The EAPOC-COPD system consists of: 1) a smart phone / tablet app or Personal Computer-based questionnaire which collects information directly from patients upon prompting, up to 1 week before their clinical appointment; and 2) a point-of-care clinical decision support system that wirelessly receives and processes questionnaire data in order to produce a symptom severity/exacerbation risk assessment, medication change recommendation, and COPD action plan, all of which is made available to providers through a prompt, upon opening the patient chart in the existing EMR. Once approved, the personalized COPD action plan is automatically populated within the patient app/portal, enabling anywhere/anytime access for patients. Patients are also provided with educational resources within their app/portal, designed to improve health literacy, inhaler technique, and adherence to their action plan
  Arms: EAPOC-COPD system
Other: Usual Care — Usual care
  Arms: Control arm

SUMMARY:
The EAPOC-COPD study is a stepped wedge cluster randomized controlled trial (SW-RCT) designed to evaluate the effectiveness of the Evidence at the Point-of-Care for COPD (EAPOC-COPD) system, a digital clinical decision support system (CDSS) integrated into primary care electronic medical records (EMRs). The system aims to improve COPD management by providing personalized pharmacotherapy recommendations, symptom and risk assessments, and self-management action plans, based on patient-reported data.

Study Design:

Six primary care sites in Ontario, Canada will transition from usual care to EAPOC-COPD-supported care in a staggered manner over 56 weeks. Each site will serve as its own control during the pre-intervention period.

Primary Objective:

To assess the impact of EAPOC-COPD on guideline-aligned pharmacotherapy optimization for COPD, measured by the proportion of patients with medication escalation.

Secondary Objectives:

Evaluate improvements in symptom/risk assessments (mMRC, CAT), COPD action plan delivery, influenza vaccination, smoking cessation support provision, pulmonary rehabilitation referrals, and COPD symptom burden

Process Measures:

Study investigators will also measure provider and patient uptake, satisfaction, and system feasibility will be assessed through EMR data audits, patient/provider surveys, and system usage analytics

Population:

All prescribers at the six primary care sites (physicians and nurse practitioners) will be eligible. The study will involve patients with physician-diagnosed COPD, identified through EMR searches.

Data Collection:

Clinical outcomes will be obtained through chart reviews and data from the Canadian Primary Care Sentinel Surveillance Network (CPCSSN), where available. Patient-reported outcomes will be captured via questionnaires through the patient app/portal.

Sample Size:

An estimated 1860 COPD patients will be seen during the study. With an expected baseline medication escalation rate of 13%, the study is powered to detect an 8% absolute increase (assuming an Intra Class Correlation (ICC) =0.1).

Analysis:

A generalized linear mixed model (GLMM) will assess primary and secondary outcomes, accounting for time trends, clustering, and the stepped roll out.

Significance:

This trial will generate real-world evidence on the effectiveness of a point-of-care digital tool in closing COPD care gaps, with potential for large-scale primary care implementation.

ELIGIBILITY:
Inclusion Criteria:

* Providers working at clinical site currently using IT infrastructure that allows for integration of EAPOC-COPD
* Providers caring for patients with COPD

Exclusion Criteria:

* Unwilling to use EAPOC-COPD system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in COPD pharmacotherapy at the provider level | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Defined by the proportion of patients whose COPD medications were escalated ("stepped-up" from short- to long-acting bronchodilator, single to dual, or dual to triple therapy), measured at the provider level

SECONDARY OUTCOMES:
Provider changes in comprehensive symptom and exacerbation risk assessment | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Will be measured by chart review, based on the presence of absence of COPD assessment test scoring
Provider changes in COPD action plan delivery | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Will be measured by chart review
Provider changes in influenza vaccination rates | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Measured by chart review
Provider changes in smoking cessation advice provision | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Measured by chart review
Provider changes in referral to pulmonary rehabilitation in appropriate patients | As provider behaviour is what is being measured, the time frame will be from site/provider recruitment (week 1) until the end of the study period (week 56)
  Measured by chart review

OTHER OUTCOMES:
Process metrics: provider uptake of EAPOC-COPD | From start of intervention period to study end at 56 weeks
  CDSS access proportion measured by system audit
Process metrics: patient uptake of EAPOC-COPD | From start of intervention period to study end at 56 weeks
  Patient questionnaire access proportion measured by system audit
User satisfaction questionnaire - providers | From week 52 to week 56 of the trial
  Questionnaires will collect demographic information and probe perceived utility of the system, readiness to adopt the system, satisfaction, and possible improvements, using open-ended and Likert scale-type questions (including the System Usability Scale - SUS)
User satisfaction questionnaire - patients | 2 weeks after first access to patient portal/app
  Questionnaires will collect demographic information and probe perceived utility of the system, readiness to adopt the system, satisfaction, and possible improvements, using open-ended and Likert scale-type questions (including the System Usability Scale - SUS)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be collecting individual patient data, but rather provider behaviour change data